CLINICAL TRIAL: NCT07159906
Title: A Phase Ib/II Prospective, Multicenter, Single-Arm Study of Homoharringtonine, BCL-2 Inhibitor, Rituximab and Prednisone in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Homoharringtonine, BCL-2 Inhibitor, Rituximab, and Prednisone in Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20250087C-R2
Record Dates: First submitted 2025-08-17; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Diffuse Large B-Cell Lymphoma; Relapsed Non-Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — Homoharringtonine; PTH2 protein, human; Lisaftoclax; Rituximab; Glucocorticoids; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HHT-Based Combination (Experimental): Patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) will receive the investigational combination of homoharringtonine, BCL2 inhibitor, rituximab, and prednisone. Treatment will be administered in 21-day cycles, with dose escalation in Phase Ib to determine dose-limiting toxicities (DLTs), maximum tolerated dose (MTD), and recommended Phase II dose (RP2D), followed by a Phase II expansion to evaluate efficacy and safety.
  Interventions: Drug: Homoharringtonine; Drug: BCL-2 inhibitor; Drug: CD20 Antibody; Drug: Glucocorticoid (GC)

INTERVENTIONS:
Drug: Homoharringtonine — A cephalotaxine alkaloid and protein synthesis inhibitor that downregulates Myeloid Cell Leukemia 1 (MCL-1), administered intravenously in 21-day cycles. Dose escalation in Phase Ib will determine dose-limiting toxicities (DLTs), maximum tolerated dose (MTD), and recommended Phase II dose (RP2D).
  Other Names: HHT
Drug: BCL-2 inhibitor — An oral selective BCL2 inhibitor administered once daily D1-7. Combined with homoharringtonine, rituximab, and prednisone in 21-day cycles.
  Other Names: Lisaftoclax; APG-2575
Drug: CD20 Antibody — An anti-CD20 monoclonal antibody administered intravenously, used in combination with chemotherapy or targeted regimens for B-cell malignancies.
  Other Names: Rituximab
Drug: Glucocorticoid (GC) — glucocorticoid , given as part of the combination regimen to enhance anti-lymphoma effect.
  Other Names: Prednisone

SUMMARY:
Diffuse large B-cell lymphoma (DLBCL) is the most common subtype of non-Hodgkin lymphoma in China and worldwide. Although standard immunochemotherapy with Rituximab, Cyclophosphamide, Doxorubicin Hydrochloride, Vincristine (Oncovin), and Prednisone (R-CHOP) achieves durable remissions in many patients, approximately 30-40% experience relapse or refractory disease with poor outcomes. Novel strategies are needed for patients who are not candidates for transplantation or who relapse after multiple lines of therapy.

Homoharringtonine (HHT) is a natural cephalotaxine alkaloid extracted from Cephalotaxus species, clinically approved in China for acute and chronic myeloid leukemias. It inhibits ribosomal protein synthesis, modulates oncogenic and epigenetic signaling pathways, and induces apoptosis through mitochondrial and stress-activated pathways. Importantly, HHT downregulates the anti-apoptotic protein Myeloid Cell Leukemia 1 (MCL-1), a critical resistance factor to B-cell lymphoma 2 (BCL-2) inhibitors. This provides a strong mechanistic rationale for combining HHT with a BCL-2 inhibitor, together with rituximab and prednisone, in relapsed/refractory DLBCL.

This prospective, multicenter, single-arm, Phase Ib/II study will evaluate the safety, tolerability, and efficacy of HHT, a BCL-2 inhibitor, rituximab, and prednisone in adult patients with relapsed/refractory DLBCL. Phase Ib will enroll 15-22 patients to determine the maximum tolerated dose (MTD), dose-limiting toxicities (DLT), and the recommended phase II dose (RP2D) of HHT. Phase II will enroll 40 patients treated at RP2D to evaluate the overall response rate (ORR) after 3 and 6 cycles per Lugano 2014 criteria. Secondary endpoints include complete remission (CR), partial remission (PR), progression-free survival (PFS), and overall survival (OS). Exploratory analyses will incorporate molecular biomarkers such as genomic profiling, circulating tumor DNA (ctDNA), and spatial transcriptomics.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, single-arm, Phase Ib/II clinical trial designed to evaluate the safety, tolerability, and efficacy of homoharringtonine (HHT), a B-cell lymphoma 2 (BCL-2) inhibitor, rituximab, and prednisone in patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL). Despite the curative potential of rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP), approximately 30-40% of patients experience relapse or refractory disease, and outcomes remain poor, especially in those not eligible for transplantation or those relapsing after multiple prior therapies.

Homoharringtonine is a cephalotaxine alkaloid approved in China for myeloid malignancies. It inhibits protein synthesis and downregulates Myeloid Cell Leukemia 1 (MCL-1), an important resistance factor to BCL-2 inhibition. Venetoclax (or Lisaftoclax, depending on study drug) is a selective oral BCL-2 inhibitor that restores apoptosis in tumor cells. Preclinical data demonstrate synergistic cytotoxicity when combining HHT with BCL-2 inhibition through complementary apoptotic mechanisms. Rituximab, an anti-CD20 monoclonal antibody, and prednisone, a glucocorticoid, further enhance anti-lymphoma activity and are established components of immunochemotherapy.

Phase Ib will use a 3+3 dose-escalation design to determine the maximum tolerated dose (MTD), dose-limiting toxicities (DLTs), and the recommended Phase II dose (RP2D) of HHT. Phase II will subsequently treat patients at the RP2D to assess overall response rate (ORR) as the primary efficacy endpoint, evaluated after 3 and 6 cycles according to Lugano 2014 criteria. Secondary endpoints include complete remission (CR), partial remission (PR), progression-free survival (PFS), overall survival (OS), and safety outcomes.

Exploratory biomarker analyses will be performed to investigate predictors of treatment response. These include targeted gene sequencing, monitoring of circulating tumor DNA (ctDNA), and spatial transcriptomic profiling in selected patients. The findings are expected to provide important insights into the clinical potential of HHT combined with BCL-2 inhibition in relapsed/refractory DLBCL, and may inform the design of biomarker-guided treatment strategies in the future.

ELIGIBILITY:
Phase II Inclusion Criteria

1. Histopathologically confirmed CD20-positive diffuse large B-cell lymphoma;
2. Age ≥18 years at enrollment, regardless of gender, with an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3;
3. Disease is refractory to or progresses within one year after first-line standard therapy containing anti-CD20 monoclonal antibodies and anthracycline-based chemotherapy, or has failed or relapsed after second-line or later standard treatment regimens, or has relapsed after autologous hematopoietic stem cell transplantation (more than 6 months post-transplant);
4. At least one measurable lesion present (as defined by the Lugano 2014 response criteria: measurable lesion is defined as a lymph node lesion with a longest diameter >1.5 cm on CT axial imaging, or an extranodal lesion with a longest diameter >1.0 cm, and 18F-FDG PET/CT positive lesion);
5. Able to provide written informed consent and capable of understanding and complying with all study requirements.

Phase II Exclusion Criteria

1. Patients with poor compliance or inability to attend regular follow-up visits;
2. Presence of severe organ dysfunction, as judged by the investigator, that renders the patient unsuitable for participation in this trial;
3. Absolute neutrophil count < 1.0 × 10⁹/L, platelet count < 50 × 10⁹/L, or hemoglobin < 80 g/L (excluding cases due to lymphoma bone marrow infiltration);
4. Other factors, as determined by the investigator, that may lead to forced early withdrawal from the study, such as other serious medical conditions (including psychiatric disorders) requiring concomitant treatment, alcoholism, drug abuse, or family/social factors that may affect patient safety or compliance;
5. History of immunodeficiency, including HIV-positive status, or other acquired or congenital immunodeficiency diseases;
6. Pregnant or breastfeeding women, and fertile patients unwilling to use contraception.
7. Acute or chronic active hepatitis B or C infection, with HBV DNA > 2000 IU/mL or 10⁴ copies/mL, or HCV RNA > 10³ copies/mL;
8. Central nervous system (CNS) metastases; however, patients with asymptomatic CNS metastases or those with symptoms that have been treated and stabilized for ≥4 weeks may be eligible;
9. Prior history of allogeneic hematopoietic stem cell transplantation;
10. Cardiac dysfunction: baseline Corrected QT interval (QTc) ≥ 500 ms; Left Ventricular Ejection Fraction (LVEF) < 45%, or New York Heart Association (NYHA) classification Class III/IV heart failure;
11. Known severe hypersensitivity to benzyl alcohol or any other components of the study drugs;
12. Requirement for concomitant use of strong CYP3A4 inducers due to medical necessity.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities (DLT) | Cycle 1 (first 21-day cycle)
  Incidence of dose-limiting toxicities assessed during Cycle 1, according to NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Maximum Tolerated Dose (MTD) | End of Phase Ib dose-escalation
  The highest dose level at which ≤1 out of 6 patients experience a DLT, determined during dose-escalation phase.
Recommended Phase II Dose (RP2D) | End of Phase Ib dose-escalation
  RP2D determined based on DLT, MTD, safety, and preliminary efficacy findings in Phase Ib.
Overall Response Rate (ORR) | At Cycle 3 and Cycle 6
  Proportion of patients achieving CR or PR, assessed per Lugano 2014 criteria using Positron Emission Tomography-Computed Tomography (PET-CT) or Computed Tomography (CT).

SECONDARY OUTCOMES:
Complete Response (CR) Rate | At Cycle 3 and Cycle 6
  Proportion of patients achieving complete response, assessed per Lugano 2014 criteria using PET-CT/CT.
Partial Response (PR) Rate | At Cycle 3 and Cycle 6
  Proportion of patients achieving partial response, assessed per Lugano 2014 criteria using PET-CT/CT.
Progression-Free Survival (PFS) | Up to 24 months from enrollment
  Time from enrollment to disease progression or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to 24 months from enrollment
  Time from enrollment to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, The First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD) outside the study group.